CLINICAL TRIAL: NCT05373875
Title: Comparison of Huntleigh Dopplex DMX Digital Doppler Arterial Waveform With the Gold Standard of Ultrasound Duplex Arterial Waveform
Status: Completed | Type: Observational
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DT/2018/6670
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Ultrasonography, Doppler; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — Doppler to listen and classify the arterial signal in the ankle and arm (Ankle brachial pressure index (ABPI))

SUMMARY:
NICE guidelines recommend an Ankle brachial pressure index (ABPI) as the primary assessment tool for patients presenting with symptoms or are at a high risk of developing peripheral arterial disease (PAD). An ABPI is typically performed using a hand-held Doppler to listen and classify the arterial signal in the ankle and arm and the systolic pressure is taken in each to create a ratio of the pressure in the ankle to the arm. New Huntleigh Dopplex DMX Digital Dopplers within the vascular department have an arterial waveform display to help interpretation of the audible signal.

This study aims to compare the audible and visual waveform traces on the Huntleigh Dopplex with the gold standard of ultrasound duplex to assess the accuracy of the trace using diagnostic measurements and the ability of clinicians to correctly identify audible and visual waveforms.

DETAILED DESCRIPTION:
A sample size of 30 patients is recommended for a pilot study to give a stable estimate of statistical parameters (mean and variance for example). Patients recruited for this study will be out patients referred for an ABPI or exercise ABPI.A participant information sheet will be sent to the patient with there invitation to book an appointment. The patient will be asked if they have read the information and if they wish to participate when they call to book an appointment. Written consent will be obtained on the day of their appointment and patients will have the opportunity to ask questions. Patients who have been admitted to hospital, have a known allergy to coupling gel, are unable to give consent, or pedal pulses are not detectable will be excluded from this study. Persons interpreting waveforms will be excluded if they reported having any hearing or visual impairment. During the appointment, each patient will be in a supine position and an 8 MHz Doppler probe from the Huntleigh Dopplex will be placed on the posterior tibial and anterior tibial arteries at the ankle of both feet applying a 45-60° angle to the surface of the skin. Audible and visual waveform traces will be recorded in each vessel on the Huntleigh Dopplex. A linear ultrasound probe from a GE 9logic will be placed on the skin in the same position as the Huntleigh Dopplex probe. The optimised spectral Doppler trace and audible waveform will be recoded on a cine loop. All recordings will be collected by the primary researcher using the same handheld Doppler and model of ultrasound machine to avoid interoperable variability. Once duplex recordings have been obtained, the patient's appointment will continue as to the department's protocol for performing an ABPI or exercise ABPI and the patient will then be discharged.

Audible and visual traces from duplex and the Huntleigh will be downloaded. Vascular trainee's in the 1st, 2nd and 3rd years of the scientist training programme and senior vascular scientists will be instructed on predefined waveforms. Audible waveforms and visual traces from the Huntleigh Dopplex will be separated and ordered randomly using a random number generator. Clinicians will listen to waveform recordings, assess visual traces and will be asked to describe them and also determine if this signifies the presence or absence of disease. Results will be analysed using descriptive statistics.

Diagnostic measurements will be taken including pulsatility and resistive index will be calculated to assess for agreement or significant difference between measurements taken on the Huntleigh Dopplex and Duplex ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Vascular Science department at University Hospitals Bristol and Weston NHS Foundation Trust for an ABPI or exercise ABPI.

Exclusion Criteria:

* Those who have been admitted to hospital,
* Under the age of 18,
* Known allergy to coupling gel,
* Unable to give consent,
* Pedal pulses are not detectable will be excluded from this study,
* Persons interpreting waveforms will be excluded if they reported having any hearing or visual impairment.

Full Set of Project Data IRAS Version 5.9.1 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Vascular Science department at University Hospitals Bristol and Weston NHS Foundation Trust ( Tertiary Care Centre)
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Change in wavefrom | 1 day
  Primary outcomes are the change in waveform identified and diagnosis of the presence or absence of disease once the visual waveform trace and assess they are sufficiently in agreement.

SECONDARY OUTCOMES:
resistive and pulsatility indexes | 1 day
  Secondary outcomes are to calculate the resistive and pulsatility indexes from the Huntleigh handheld Dopplex and duplex ultrasound arterial waveforms and assess if they are sufficiently in agreement

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Robinson, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (1):
- University Hospitals Bristol and Weston NHS Foundation Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No